CLINICAL TRIAL: NCT02780661
Title: A Method Development Clinical Study to Investigate the Efficacy of the Different Frequencies of Use of a Denture Cleanser
Brief Title: Frequency of Denture Cleanser Use and Denture Cleanliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 205202
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Denture Cleansers
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Denture Cleanser Daily Use Period (Experimental): Participants will be instructed to soak upper arch dentures in the evening in cup of very warm water (150 millilitre [ml]) with 1 denture cleansing tablet from Day 0 to Day 7 for 15 minutes (mins). Brush dentures for 30 seconds using the solution, rinse under running water for 10 seconds. Cleaning of upper arch dentures in the morning is not permitted. Lower arch dentures will be cleaned using the participant's normal oral hygiene procedures in the morning and evening. If the participants will have lower removable partial or complete dentures, the soaking of these dentures will be done in a separate cup from the cup provided for soaking the upper denture.
  Interventions: Device: Denture Cleanser Daily Use Period; Other: Water
- Denture Cleanser Weekly Use Period (Experimental): Participants will be instructed to soak upper arch dentures in the evening in cup of very warm water (150 ml) from Day 0 to Day 6 for 15 mins; and in cup of very warm water (150 ml) with 1 denture cleansing tablet on Day 7 at site for 15 mins. Brush dentures for 30 seconds using the solution, rinse under running water for 10 seconds. Cleaning of upper arch dentures in the morning is not permitted. Lower arch dentures will be cleaned using the participant's normal oral hygiene procedures in the morning and evening. If the participants will have lower removable partial or complete dentures, the soaking of these dentures will be done in a separate cup from the cup provided for soaking the upper denture.
  Interventions: Device: Denture Cleanser Weekly Use Period; Other: Water

INTERVENTIONS:
Device: Denture Cleanser Daily Use Period — One denture cleansing tablet will be soaked in a cup of very warm water (150 ml) with dentures for Day 0 to Day 7 for 15 mins. Brush dentures for 30 seconds using the solution, rinse under running water for 10 seconds.
  Other Names: Corega tablet
  Arms: Denture Cleanser Daily Use Period
Device: Denture Cleanser Weekly Use Period — One denture cleansing tablet will be soaked in cup of very warm water (150 ml) from Day 0 to Day 6 for 15 mins; and in cup of very warm water (150 ml) with 1 denture cleansing tablet on Day 7 at site for 15 mins. Brush dentures for 30 seconds using the solution, rinse under running water for 10 seconds.
  Other Names: Corega tablet
  Arms: Denture Cleanser Weekly Use Period
Other: Water — A cup of very warm water will be used to soak one denture cleansing tablet and dentures for per day (Day 0 to Day 7) or weekly (Day 0 and Day 7) treatment regimen.

SUMMARY:
This method development study will be a two treatment arm, randomized, cross over study in a population with edentulous upper arch restored with a maxillary complete denture. The lower may be a partial or full edentulous mandibular arch that may be restored with a stable complete, partial or implant supported denture.

DETAILED DESCRIPTION:
This is a single-center, 2 treatment periods, examiner-blind, randomized, 7 day crossover study in adult participants with a complete maxillary denture. This is a method development study to investigate the changes in the level of denture plaque, microbial counts, microbial composition and stain on the maxillary dentures after daily denture cleanser use versus dentures that are cleaned weekly.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged between 18 and 84 years inclusive.
* Good general and mental health with, in the opinion of the Investigator or medically qualified designee: No clinically significant and relevant abnormalities in medical history or upon oral examination; Absence of any condition that could affect the participant's safety or wellbeing or their ability to understand and follow study procedures and requirements.
* Maxillary Arch: Completely edentulous maxillary arch restored with a conventional full acrylic based upper complete denture.
* Mandibular Arch: Dentate, partial or full edentulous mandibular arch. Partial or full edentulous arch may be restored with a stable complete, partial or implant supported denture. (Mandibular dentures are not used for assessments or measures).
* Maxillary dentures must be considered to be moderately well-fitting at the screening visit. (Kapur Index, Olshan Modification: retention score >2, stability score >2).
* Maxillary dentures must be considered to be well-made based on design and construction criteria specified in the protocol.

Exclusion Criteria:

* Women who are breast-feeding, are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Previous participation in this study or in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.
* Recent history (within the last year) of alcohol or other substance abuse.
* Current or relevant history of any serious, severe or unstable physical or psychiatric illness or any other medical condition (e.g. Diabetes Mellitus) that would make the participant unlikely to fully complete the study or any that increases the risk to the participant or undermines the data validity.
* Implanted with a cardiac pacemaker.
* Daily doses of medication (example Antibiotics, Inhaled steroids etc.) that might interfere with ability to perform the study according to protocol or might affect the efficacy assessments (as determined by the Investigator/ Examiner).
* Any clinically significant or relevant oral abnormality that, in the opinion of the Investigator, could affect the participant's participation in the study.
* Any pre-existing oral irritations.
* Any recent (within 30 days) gingival /oral surgery.
* Participants who are unwilling to refrain from smoking, including e-cigarettes and the use of chewing tobacco or other tobacco products for the duration of the study.
* An employee of the sponsor or the study site or members of their immediate family.
* An employee of any toothpaste manufacturer or their immediate family.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Glasgow, United Kingdom

REFERENCES:
- [Derived] Ramage G, O'Donnell L, Sherry L, Culshaw S, Bagg J, Czesnikiewicz-Guzik M, Brown C, McKenzie D, Cross L, MacInnes A, Bradshaw D, Varghese R, Gomez Pereira P, Jose A, Sanyal S, Robertson D. Impact of frequency of denture cleaning on microbial and clinical parameters - a bench to chairside approach. J Oral Microbiol. 2018 Oct 29;11(1):1538437. doi: 10.1080/20002297.2018.1538437. eCollection 2019. PMID 30598732
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=205202&attachmentIdentifier=0421ade3-f0ca-4bd9-a65e-579addc40b8e&fileName=gsk-205202-reporting-and-analysis-plan-redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=205202&attachmentIdentifier=853435c5-a924-4e84-9905-c35ea584a25e&fileName=gsk-205202-protocol-redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=205202&attachmentIdentifier=d973323e-85c6-4535-b022-4d76ad9842c5&fileName=gsk-205202-clinical-study-report-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at a single center in United Kingdom.
Pre-assignment Details: A total of 25 participants were screened, out of which 19 participants were randomized to the study, 6 participants were not randomized because of screening failure.
Groups:
- Denture Cleanser Tablet: Daily Use /Weekly Use: Participants were instructed to soak upper arch dentures in cup of very warm water (150 milliliter [mL]) with 1 denture cleansing tablet from Day 0 to Day 7 for 15 minutes (min.) (supervised product use at site: Day 0,3,7; home use of product in evening for rest of days) in treatment period 1. Following 7 day wash out period, same participants were instructed to soak upper arch dentures in cup of very warm water (150 mL) from Day 0 to Day 6 for 15 mins (supervised product use at site: Day 0,3; home use of product in evening for rest of days); and in cup of very warm water (150 mL) with 1 denture cleansing tablet on Day 7 at site for 15 mins in treatment period 2. Participants were also instructed to brush dentures for 30 seconds using solution, rinse under running water for 10 seconds during each treatment period. Cleaning of upper arch dentures in morning was not permitted. Lower arch dentures were cleaned using participant's normal oral hygiene procedures in morning & evening.
- Denture Cleanser Tablet: Weekly Use/ Daily Use: Participants were instructed to soak upper arch dentures in cup of very warm water (150 mL) from Day 0 to Day 6 for 15 mins (supervised product use at site: Day 0,3; home use of product in evening for rest of days) and in cup of very warm water (150 mL) with 1 denture cleansing tablet on Day 7 at site for 15 mins in treatment period 1. Following 7 day wash out period, same participants were instructed to soak upper arch dentures in cup of very warm water (150 mL) with 1 denture cleansing tablet from Day 0 to Day 7 for 15 minutes (min.) (supervised product use at site: Day 0,3,7; home use of product in evening for rest of the days) in treatment period 1. Participants were also instructed to brush dentures for 30 seconds using solution, rinse under running water for 10 seconds during each treatment period. Cleaning of upper arch dentures in morning was not permitted. Lower arch dentures were cleaned using participant's normal oral hygiene procedures in morning & evening.
Period: Period 1
Arm/Group | Denture Cleanser Tablet: Daily Use /Weekly Use | Denture Cleanser Tablet: Weekly Use/ Daily Use
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Wash Out Period
Arm/Group | Denture Cleanser Tablet: Daily Use /Weekly Use | Denture Cleanser Tablet: Weekly Use/ Daily Use
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Denture Cleanser Tablet: Daily Use /Weekly Use | Denture Cleanser Tablet: Weekly Use/ Daily Use
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were included for baseline evaluation.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (5.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 19
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Aerobic Bacteria Microbial Count on Day 7
Description: Microbial count samples were collected using a paper disc (disc sampling). A pre-sterilised 10-millimeter (mm) filter paper disc was lightly pressed against the selected quadrant of maxillary denture, leaving enough space to place two discs without overlap. The selected areas were lateral to the midline and corresponding to the palatal rugae. Microbiological sampling was carried out from one standardised site on the fitting surface of the denture for standard culture. The discs were left for 20 secs prior to aseptic removal using sterile tweezers, and were serially diluted and plated into appropriate agar plates and incubated aerobically. Pre-treatment samples were taken from the left rough and left smooth denture surface. Post-treatment samples were taken from the right rough and right smooth denture surface at Day 7.
Time Frame: Baseline (Day 0 pre-treatment), Day 7 (post-treatment)
Population: Analysis for this outcome was performed on intent-to-treat (ITT) population which included all participants who were randomized, received at least one dose of the study treatment and provided at least one post-baseline assessment of microbial count from disc sampling.
Measure: Mean (Standard Deviation); unit: log10(CFU[colony forming unit]/disc+1)
Groups:
- Denture Cleanser Tablet: Daily Use Period: Participants were instructed to soak upper arch dentures in cup of very warm water (150 mL) with 1 denture cleansing tablet from Day 0 to Day 7 for 15 min. (supervised product use at site: Day 0,3,7; home use of product in evening for rest of days). Participants were also instructed to brush dentures for 30 seconds using solution, rinse under running water for 10 seconds during each treatment period. Cleaning of upper arch dentures in morning was not permitted. Lower arch dentures were cleaned using participant's normal oral hygiene procedures in morning & evening.
- Denture Cleanser Tablet: Weekly Use: Participants were instructed to soak upper arch dentures in cup of very warm water (150 mL) from Day 0 to Day 6 for 15 mins (supervised product use at site: Day 0,3; home use of product in evening for rest of days) and in cup of very warm water (150 mL) with 1 denture cleansing tablet on Day 7 at site for 15 mins. Participants were also instructed to brush dentures for 30 seconds using solution, rinse under running water for 10 seconds during each treatment period. Cleaning of upper arch dentures in morning was not permitted. Lower arch dentures were cleaned using participant's normal oral hygiene procedures in morning & evening.
Arm/Group | Denture Cleanser Tablet: Daily Use Period | Denture Cleanser Tablet: Weekly Use
Number analyzed (Participants) | 19 | 19
log10(CFU[colony forming unit]/disc+1) | -1.78 (2.248) | -1.20 (2.636)
Statistical Analysis 1: Comparison: Denture Cleanser Tablet: Daily Use Period vs Denture Cleanser Tablet: Weekly Use; H0: There is no treatment difference between daily and weekly product use. H1: There is a treatment difference between daily and weekly product use; Test type: Other; p = 0.0144, ANCOVA — Log10 change from baseline in aerobic bacteria microbial count as response variable, treatment and period as fixed effect, participant level and period level pre-treatment microbial count as covariates and participant as random effect; Least square (LS) mean difference = -0.86, 95% CI 2-sided [-1.530 to -0.196] — Difference is first named treatment minus second named treatment in log10{(count+1)/(baseline+1)} such that a negative difference favors the first named treatment

2. Primary Outcome: Change From Baseline in Anaerobic Bacteria Microbial Count on Day 7
Description: Microbial count samples were collected using a paper disc (disc sampling). A pre-sterilised 10 mm filter paper disc was lightly pressed against the selected quadrant of maxillary denture, leaving enough space to place two discs without overlap. The selected areas were lateral to the midline and corresponding to the palatal rugae. Microbiological sampling was carried out from one standardised site on the fitting surface of the denture for standard culture. The discs were left for 20 secs prior to aseptic removal using sterile tweezers, and were serially diluted and plated into appropriate agar plates and incubated anaerobically. Pre-treatment samples were taken from the left rough and left smooth denture surface. Post-treatment samples were taken from the right rough and right smooth denture surface at Day 7.
Time Frame: Baseline (Day 0 pre-treatment), Day 7 (post-treatment)
Population: ITT Population defined as all participants who are randomized, received at least one dose of study treatment and have at least one post-baseline assessment of microbial count from disc sampling.
Measure: Mean (Standard Deviation); unit: log10(CFU/disc+1)
Groups:
- Denture Cleanser Tablet: Daily Use: Participants were instructed to soak upper arch dentures in cup of very warm water (150 mL) with 1 denture cleansing tablet from Day 0 to Day 7 for 15 min. (supervised product use at site: Day 0,3,7; home use of product in evening for rest of days). Participants were also instructed to brush dentures for 30 seconds using solution, rinse under running water for 10 seconds during each treatment period. Cleaning of upper arch dentures in morning was not permitted. Lower arch dentures were cleaned using participant's normal oral hygiene procedures in morning & evening.
Arm/Group | Denture Cleanser Tablet: Daily Use | Denture Cleanser Tablet: Weekly Use
Number analyzed (Participants) | 19 | 19
log10(CFU/disc+1) | -1.57 (2.478) | -1.54 (2.586)
Statistical Analysis 1: Comparison: Denture Cleanser Tablet: Daily Use vs Denture Cleanser Tablet: Weekly Use; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.1879, ANCOVA — Log10 change from baseline in anaerobic bacteria microbial count as response variable, treatment and period as fixed effect, participant level and period level pre-treatment microbial count as covariates and participant as random effect; LS mean difference = -0.48, 95% CI 2-sided [-1.230 to 0.261] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Change From Baseline in Candidal Microbial Count on Day 7
Description: Microbial count samples were collected using a paper disc (disc sampling). A pre-sterilised 10 mm filter paper disc was lightly pressed against the selected quadrant of maxillary denture, leaving enough space to place two discs without overlap. The selected areas were lateral to the midline and corresponding to the palatal rugae. Microbiological sampling was carried out from one standardised site on the fitting surface of the denture for standard culture. The discs were left for 20 secs prior to aseptic removal using sterile tweezers, and were serially diluted and plated into appropriate agar plates and incubated aerobically. Pre-treatment samples were taken from the left rough and left smooth denture surface. Post-treatment samples were taken from the right rough and right smooth denture surface at Day 7.
Time Frame: Baseline (Day 0 pre-treatment), Day 7 (post-treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10(CFU/disc+1)
Arm/Group | Denture Cleanser Tablet: Daily Use | Denture Cleanser Tablet: Weekly Use
Number analyzed (Participants) | 19 | 19
log10(CFU/disc+1) | 0.0 (0.0) | 0.0 (0.0)

4. Secondary Outcome: Change From Baseline in Aerobic Bacteria Microbial Count on Day 3
Description: Microbial count samples were collected using a paper disc (disc sampling). A pre-sterilised 10 mm filter paper disc was lightly pressed against the selected quadrant of maxillary denture, leaving enough space to place two discs without overlap. The selected areas were lateral to the midline and corresponding to the palatal rugae. Microbiological sampling was carried out from one standardised site on the fitting surface of the denture for standard culture. The discs were left for 20 secs prior to aseptic removal using sterile tweezers, and were serially diluted and plated into appropriate agar plates and incubated aerobically. Pre-treatment samples were taken from the left rough and left smooth denture surface. Post-treatment samples were taken from the right rough and right smooth denture surface at Day 3.
Time Frame: Baseline (Day 0 pre-treatment), Day 3 (post-treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10(CFU/disc+1)
Arm/Group | Denture Cleanser Tablet: Daily Use | Denture Cleanser Tablet: Weekly Use
Number analyzed (Participants) | 19 | 19
log10(CFU/disc+1) | -1.74 (1.917) | 0.36 (3.019)

5. Secondary Outcome: Change From Baseline in Anaerobic Bacteria Microbial Count on Day 3
Description: Microbial count samples were collected using a paper disc (disc sampling). A pre-sterilised 10 mm filter paper disc was lightly pressed against the selected quadrant of maxillary denture, leaving enough space to place two discs without overlap. The selected areas were lateral to the midline and corresponding to the palatal rugae. Microbiological sampling was carried out from one standardised site on the fitting surface of the denture for standard culture. The discs were left for 20 secs prior to aseptic removal using sterile tweezers, and were serially diluted and plated into appropriate agar plates and incubated anaerobically. Pre-treatment samples were taken from the left rough and left smooth denture surface. Post-treatment samples were taken from the right rough and right smooth denture surface at Day 3.
Time Frame: Baseline (Day 0 pre-treatment), Day 3 (post-treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10(CFU/disc+1)
Arm/Group | Denture Cleanser Tablet: Daily Use | Denture Cleanser Tablet: Weekly Use
Number analyzed (Participants) | 19 | 19
log10(CFU/disc+1) | -1.74 (2.134) | 1.08 (2.753)

6. Secondary Outcome: Change From Baseline in Candidal Microbial Count on Day 3
Description: as for outcome 4
Time Frame: Baseline (Day 0 pre-treatment), Day 3 (post-treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10(CFU/disc+1)
Arm/Group | Denture Cleanser Tablet: Daily Use | Denture Cleanser Tablet: Weekly Use
Number analyzed (Participants) | 19 | 19
log10(CFU/disc+1) | 0.0 (0.0) | 0.0 (0.0)

ADVERSE EVENTS:
Time Frame: up to 31 days (from the start of denture and dental prophylaxis at the Screening Visit until 5 days following last administration of the study product at Visit 8)
Arm/Group | Denture Cleanser Tablet: Daily Use | Denture Cleanser Tablet: Weekly Use
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 8/19 | 8/19
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Denture Cleanser Tablet: Daily Use (N=19) | Denture Cleanser Tablet: Weekly Use (N=19)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral mucosal erythema (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tongue coated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injury associated with device (General disorders) | 4 (4) | 3 (4)
Chronic fatigue syndrome (General disorders) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.